CLINICAL TRIAL: NCT00037739
Title: Chronic Obstructive Pulmonary Disease Gene Localization
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1175; R01HL067469 (NIH)
Record Dates: First submitted 2002-05-20; First posted 2002-05-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Lung Diseases; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To localize within the genome a chronic obstructive pulmonary disease susceptibility gene.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease (COPD) is a slowly progressive disorder characterized by airways obstruction that lasts for at least several months. The two major causes of COPD are chronic bronchitis and emphysema. Either disorder may occur with or without airways obstruction, but airways obstruction causes impairment of lung function leading to disability and death. COPD is a major health problem in the United States and throughout the world, consistently ranking among the most common causes of death in the United States. Cigarette smoking is the primary environmental factor that increases the risk of COPD, but other environmental factors have also been implicated. However, despite a well-established role, environmental factors alone do not cause COPD. Symptomatic COPD develops in only 10-20 percent of heavy cigarette smokers, probably those with a genetic susceptibility, although common COPD susceptibility genes have yet to be identified.

DESIGN NARRATIVE:

The study applied statistical linkage analysis to family data. Pulmonary measurements had already been collected on 159 members of 16 pedigrees and evidence supporting a COPD susceptibility gene in these pedigrees had been obtained from segregation analysis. Each of 11,995 genetic markers, which had already been genotyped on pedigree members, were tested for evidence of linkage to the inferred COPD susceptibility gene. Evidence of linkage to one or more genetic markers identifed genomic locations of COPD susceptibility genes. The high density of markers allowed fine-mapping of the gene. Successful completion of this gene localization project was the necessary prerequisite for a project to identify and characterize a COPD susceptibility gene. Identifying a gene that when mutated increased the risk of COPD may increase understanding of pulmonary function, as well as allowing gene-carriers to be identified and made aware of their susceptibility.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Hasstedt — University of Utah

REFERENCES:
- [Background] Malhotra A, Peiffer AP, Ryujin DT, Elsner T, Kanner RE, Leppert MF, Hasstedt SJ. Further evidence for the role of genes on chromosome 2 and chromosome 5 in the inheritance of pulmonary function. Am J Respir Crit Care Med. 2003 Sep 1;168(5):556-61. doi: 10.1164/rccm.200303-410OC. Epub 2003 Jun 5. PMID 12791583
- [Background] Malhotra A, Cromer K, Leppert MF, Hasstedt SJ. The power to detect genetic linkage for quantitative traits in the Utah CEPH pedigrees. J Hum Genet. 2005;50(2):69-75. doi: 10.1007/s10038-004-0222-8. Epub 2005 Jan 29. PMID 15682273